CLINICAL TRIAL: NCT05286996
Title: Cryoneurolysis for Pain Management After Total Knee Arthroplasty - a Pilot Study
Brief Title: Cryoneurolysis for TKA - a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-iovera
Record Dates: First submitted 2022-03-01; First posted 2022-03-18 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Knee Pain Chronic; Osteoarthritis
Keywords: total knee artroplasty; knee replacement
MeSH Terms: conditions — Osteoarthritis | interventions — Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: Parallel-randomized participant-blinded control trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes assessors will be blinded about treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iovera (Experimental): Cryoneurolysis + standard of care: Usual intervention plus pre-operation Iovera treatment. Patients will receive local anaesthesia unilaterally to the affected knee prior to the treatment and then the anesthesiologist will administer the freezing cold therapy (Iovera device) to the affected knee.
  Interventions: Device: Iovera - Cryoneurolysis
- Placebo (Placebo Comparator): Placebo: Usual intervention plus pre-operation placebo. The placebo group will receive short-acting local anaesthesia injection unilaterally to the affected knee.
  Interventions: Drug: Local anesthetic

INTERVENTIONS:
Device: Iovera - Cryoneurolysis — Iovera system delivers precise, controlled doses of cold temperature only to the targeted nerve through a handheld device.
  Arms: Iovera
Drug: Local anesthetic — Placebo - local anaesthesia
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Total Knee Arthroplasty (TKA) is also known as a knee replacement. It is one of the most common orthopaedic (bone) surgeries performed and is usually very successful, but some people who have had a knee replacement feel pain that lasts for at least 3 months after surgery and thus continue to take pain control/ analgesic (opioids) medication. Opiates are medications like morphine.

Pain post-surgery can make it difficult to recover and return to daily activities. A better control of pain before the surgery, can help people feel less pain, recover faster, and use less opioids after surgery.

Cryoneurolysis means freezing the nerves that can cause pain. It uses very low temperatures in a specific body part (e.g., nerves to the knee) to freeze the pain nerves and therefore reduce the pain. When applied before the surgery it might help with postoperative pain after knee replacement.

This study will evaluate Iovera, a cryoneurolysis handheld device commercially available in Canada that delivers freezing cold to a target nerve by using nitrous oxide. Cryoneurolysis can relieve pain and symptoms associated with osteoarthritis of the knee for up to 90 days.

DETAILED DESCRIPTION:
Patients undergoing total knee replacement (TKA) often experience a significant amount of pain during the immediate postoperative period, thus appropriate pain management before, during and after the surgery is a key component of patient satisfaction and better outcomes.

Opioids are the most commonly prescribed drugs to manage postoperative orthopaedic pain; however, their well-known side effects, such as nausea, vomiting and the potential high risk for dependence, can slow down recovery and lead to substance disorders.

Studies have reported, that more than 20% of patients receiving TKA experience persistent and unchanged pain post-surgery. Moreover, 15 to 25% of TKA patients continue the use of opioids at 3 months after surgery, 35% of patients report pain that interferes with their activities of daily living 4 months after surgery.

Adequate pain management before the surgery may prevent or reduce the rate of persistent pain and opioid usage after TKA. Cryoneurolysis is a minimally invasive procedure that uses a small probe to freeze [at very low temperatures - below -20oC] the target nerve. It can promote regeneration of the structure and function of the affected nerve. It has shown promising short and long-term results in a variety of acute and chronic pain conditions.

Retrospective studies revealed that preoperative cryoneurolysis might be efficacious in attenuating pain improving function and reducing opioid prescription 12 weeks after TKA. However, the studies are mostly retrospective, with small numbers of patients and not standardized knee specific outcomes.

This is a pilot randomized clinical trial to establish the feasibility of administering the study device (Iovera) to our target population as well as to test and refine the recruitment criteria, study design, patient acceptability, and operational strategies for use in a large definitive study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* 18 to 80 years of age
* Patients with radiographic confirmation and clinical correlation for severe osteoarthritis diagnosis with an indication for total knee replacement
* Patients undergoing primary unilateral total knee replacement
* No previous unilateral knee injection (steroids/biologics) within 6 months of study
* The patient is able to read and understand English and provide informed consent to participation in the study

Exclusion Criteria:

* Pregnancy and breastfeeding
* Cryoglobulinemia
* Paroxysmal cold hemoglobinuria
* Cold urticaria
* Raynaud's disease
* Current Opioid use
* History of opiate, narcotic and alcohol abuse
* Revision total knee replacement surgery
* Open and/or infected wounds at or near the affected knee

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient recruitment rate | 12 months postoperative
  The primary objective of the pilot trial is to establish the feasibility of a larger definitive trial by successfully recruiting 20 patients over a 12-month period.

SECONDARY OUTCOMES:
Opioid consumption | 2 weeks postoperative
  Cumulative opioid consumption will be assessed by drug diaries that patients will bring back to the hospital visit at 2 week follow up appointment.
Numeric Rating Scale of Pain | 2, 6 and 12 weeks postoperative
  It consists of 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme.
Oxford Knee score | 6 and 12 weeks postoperative
  is a validated 12-item patient-reported outcome specifically designed and developed to assess function and pain after total knee replacement surgery. It scores from 0 (might indicate severe arthritis) to 48 (normal joint function).
EQ-5D-5L | 6 and 12 weeks postoperative
  It is a health-related quality of life measure that consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ-VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ-VAS records the patient's self-rated health on a vertical visual analogue scale.
Quality of Recovery | 12 weeks postoperative
  The 15-item Quality of Recovery (QoR-15) scale is a validated, simple, reliable, multidimensional questionnaire that measures the quality of recovery after surgery. Fifteen questions assess five domains of patient-reported health status: pain, physical comfort, physical independence, psychological support and emotional state.

CONTACTS AND LOCATIONS:
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan M, Osman K, Green G, Haddad FS. The epidemiology of failure in total knee arthroplasty: avoiding your next revision. Bone Joint J. 2016 Jan;98-B(1 Suppl A):105-12. doi: 10.1302/0301-620X.98B1.36293. PMID 26733654
- [Background] Choi YJ, Ra HJ. Patient Satisfaction after Total Knee Arthroplasty. Knee Surg Relat Res. 2016 Mar;28(1):1-15. doi: 10.5792/ksrr.2016.28.1.1. Epub 2016 Feb 29. PMID 26955608
- [Background] Hamilton DF, Lane JV, Gaston P, Patton JT, Macdonald D, Simpson AH, Howie CR. What determines patient satisfaction with surgery? A prospective cohort study of 4709 patients following total joint replacement. BMJ Open. 2013 Apr 9;3(4):e002525. doi: 10.1136/bmjopen-2012-002525. Print 2013. PMID 23575998
- [Background] Wylde V, Hewlett S, Learmonth ID, Dieppe P. Persistent pain after joint replacement: prevalence, sensory qualities, and postoperative determinants. Pain. 2011 Mar;152(3):566-572. doi: 10.1016/j.pain.2010.11.023. Epub 2011 Jan 15. PMID 21239114
- [Background] Zhou L, Kambin P, Casey KF, Bonner FJ, O'Brien E, Shao Z, Ou S. Mechanism research of cryoanalgesia. Neurol Res. 1995 Aug;17(4):307-11. doi: 10.1080/01616412.1995.11740333. PMID 7477749
- [Background] Zhou L, Shao Z, Ou S. Cryoanalgesia: electrophysiology at different temperatures. Cryobiology. 2003 Feb;46(1):26-32. doi: 10.1016/s0011-2240(02)00160-8. PMID 12623025
- [Background] Radnovich R, Scott D, Patel AT, Olson R, Dasa V, Segal N, Lane NE, Shrock K, Naranjo J, Darr K, Surowitz R, Choo J, Valadie A, Harrell R, Wei N, Metyas S. Cryoneurolysis to treat the pain and symptoms of knee osteoarthritis: a multicenter, randomized, double-blind, sham-controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1247-1256. doi: 10.1016/j.joca.2017.03.006. Epub 2017 Mar 20. PMID 28336454